CLINICAL TRIAL: NCT02303210
Title: Evaluation of Frequency Lowering Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 012FrL2612901
Record Dates: First submitted 2014-11-03; First posted 2014-11-27 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- hearing aid NaidaUP (Other): Within subject design: compare frequency lowering one with frequency lowering two.
  Interventions: Device: hearing aid NaidaUP
- hearing aid NaidaSP (Other): Within subject design: compare frequency lowering one with frequency lowering two.
  Interventions: Device: hearing aid NaidaSP

INTERVENTIONS:
Device: hearing aid NaidaUP — Standard Power Hearing instruments including different frequency lowering techniques
  Arms: hearing aid NaidaUP
Device: hearing aid NaidaSP — Standard Power Hearing instruments including different frequency lowering techniques
  Arms: hearing aid NaidaSP

SUMMARY:
The purpose of this study is to examine two frequency lowering techniques in case of audibility, recognition, distinction, discriminability and sound quality.

DETAILED DESCRIPTION:
This is a controlled, single blinded and randomised comparative study which is conducted monocentric at Hoerzentrum Oldenburg, Germany. The focus is to test two frequency lowering techniques with an amount of 30 moderate to severe, symmetrically sensorineural hearing impaired adult subjects. The subjects, all of them native German speakers, individually conduct a number of laboratory standard tests and home trials (questionnaires) during 6 months including seven appointments of 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* female and male adults (>18 years old)
* mild to severe Hearing Loss
* symmetric Hearing Loss
* german native speakers

Exclusion Criteria:

* persons who are not able to attend multiple appointments
* persons who are not able to handle a hearing aid
* persons with a mental handicap
* persons with limited access to multiple hearing situations
* persons with psychological disease
* no acclimatization to hearing aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Audibility improvement (Delta of dB SPL thresholds) of high frequency sounds measured with a Phoneme Perception Test. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rehmann, B.Sc., Study Chair — Phonak AG
Locations (1):
- Hoerzentrum Oldenburg, Oldenburg, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
National Regulations do not require to share data,